CLINICAL TRIAL: NCT01187030
Title: Appropriateness of Frozen Plasma Use in Canada
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Blood Services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200766101
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Blood Component Transfusion
Keywords: Frozen Plasma; Fresh Frozen Plasma; Prothrombin Complex Concentrates; RAND UCLA; Modified Delphi Methodology; Expert Panel; Appropriateness Rating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is little evidence to guide the current use of Frozen Plasma. Despite this, over 260,000 units of frozen plasma are transfused in Canada annually. Based on the limited published data available, the pattern of practice for Frozen Plasma transfusions is highly variable and an important number of Frozen Plasma transfusions appear to be inappropriate. Given inappropriate use, it is inevitable that a percentage of patients experience unnecessary and potentially life-threatening adverse transfusion reactions. Current guidelines for Frozen Plasma offer little help in guiding specific clinical decisions as their recommendations lack sufficient clinical details. This lack of detail also hinders the utility of these guidelines to help monitor and improve clinical practice. Further research examining Frozen Plasma transfusions including an understanding our current use is critical to improve the utilization of this valuable and limited resource.

DETAILED DESCRIPTION:
Objectives: We will (1) systematically review the evidence for the use of Frozen Plasma transfusions, (2) establish appropriateness ratings for all clinical scenarios for which Frozen Plasma is transfused, and (3) perform a 3-month prospective study to understand the current use and the appropriateness of use of Frozen Plasma in 12 Canadian academic centres.

Methods and Analysis: Following a well established methodology to evaluate medical therapies developed at RAND/UCLA, the investigators will purposively employ different epidemiologic techniques to assess the current use and appropriateness of Frozen Plasma transfusions in Canada.

First, we will undertake a thorough systematic review of the evidence for the use of Frozen Plasma across all indications.

The RAND modified Delphi methodology will then be used to determine the appropriateness of transfusing Frozen Plasma across a comprehensive set of clinical scenarios. A panel of 9 experts representing relevant clinical specialties will use the evidence from the systematic review to determine the appropriateness ratings (an ordinal scale of 1-9) for each clinical scenario.

Subsequently, we will undertake a prospective cohort study of all episodes of Frozen Plasma transfusions (approximately 5000 episodes) at 10 Canadian academic centres (17 hospitals) using the appropriateness ratings. Trained research assistants will identify all transfusion episodes via the blood bank and perform a chart review to obtain demographic variables (age, sex, weight), clinical variables (diagnosis, coagulopathy, indications for frozen plasma transfusions, other blood product transfusions), and laboratory (pre and posttransfusion coagulation tests) information. These data will allow mapping of each transfusion event onto a specific clinical scenario rated by the expert panel and the assignment of an appropriateness rating. We will also determine the total number of patients and the number of patients for each of the largest user groups of Frozen Plasma at each hospital. The primary outcomes for the prospective cohort study, the proportion of inappropriate transfusions (appropriateness) and the proportion of patients transfused (overall utilization), will be initially examined using descriptive statistics. Using hierarchical modeling, a logistic regression analysis will be used to examine the proportion of inappropriate transfusions while controlling for indication, hospital, and patient factors. For the analysis of overall utilization of Frozen Plasma, a chi-square analysis will be used to compare the proportion of patients transfused in the largest user groups at the different hospitals. A secondary analysis will examine the dose of Frozen Plasma transfused.

Generated Research: From the systematic reviews, appropriateness ratings, and the results of the cohort study, we will have summarized the evidence supporting the use of Frozen Plasma, produced detailed clinical guidelines outlining the appropriate and inappropriate indications for Frozen Plasma and provided an understanding of the variation in use and appropriateness of Frozen Plasma. Each of these elements can then be used by hospitals in Canada and elsewhere to improve the current use of Frozen Plasma. Understanding of the variation in Frozen Plasma will allow for a framework to improve transfusion practice and identify those areas of Frozen Plasma use that merit the greatest attention for further research.

ELIGIBILITY:
Inclusion Criteria:

* All subjects receiving frozen plasma or PCC transfusions

Exclusion Criteria:

No subjects excluded -

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at 10 academic medical centres (17 hospitals) across Canada
Sampling Method: Non-Probability Sample
Enrollment: 2580 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the appropriateness of Frozen Plasma transfusions will be the proportion of appropriate transfusion episodes. | 2 months
  Each transfusion episode will be the unit of analysis as a single patient may receive both inappropriate and appropriate transfusions.

SECONDARY OUTCOMES:
The number of units transfused per patient will be the secondary outcome. | 2 months
  The investigators consider whether or not a patient received either Frozen Plasma or a prothrombin complex concentrate as the most clinically important outcome. The investigators will also collect data on the total number of patients in hospital for the study period. This outcome is also important as differences in transfusion dose will have an important impact on the cost of Frozen Plasma and prothrombin complex concentrate transfusions and will not be captured in an analysis looking solely at the proportion of patients transfused

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Tinmouth, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute